CLINICAL TRIAL: NCT02422290
Title: Ketamine Treatment for Pediatric-Refractory Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Pablo H. Goldberg, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #7023
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Ketamine; Glutamate; OCD treatment; OCD medication
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adolescents and young adults with OCD (Experimental): All participants will be receive the intravenous ketamine infusion.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Single infusion of IV Ketamine, 0.5mg/kg
  Other Names: Ketalar

SUMMARY:
This pilot study is proposed to determine the acceptability, feasibility and potential efficacy of ketamine, a medication that modulates glutamate in the brain, as a rapid treatment for obsessive-compulsive disorder (OCD) symptoms in adolescents and young adults with OCD. This study will recruit 6 youth (ages 14-22) who are diagnosed with clinically significant OCD and have failed at least one adequate trial of a Serotonin Reuptake Inhibitor (SRI) medication and a course of Cognitive-Behavioral Therapy (CBT) (unless unable to access or tolerate) for OCD in the past. Participants will receive a single infusion of intravenous ketamine and be assessed at regular intervals post-infusion for up to 14 days. At the end of the 14-day treatment phase, all participants will be offered three months of open treatment for OCD with medication and/or CBT.

DETAILED DESCRIPTION:
See Brief Summary for description.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 14-22 years of age at the time of consent (post-pubertal)
2. Participant and a parent/guardian must be able to read and understand English
3. Participant must be physically healthy and weigh at least 25kg. If female, must not be pregnant.
4. Participant must fulfill DSM-V criteria for OCD, OCD being the principal disorder (i.e., currently the most severe and in need of treatment) and have had OCD for at least six months.
5. Participant must score ≥ 16 on the Children's Yale-Brown Obsessive Compulsive Scale (CYBOCS) prior to entering the study, report at least moderate severity of obsessions and/or compulsions..
6. Participant must have tried and failed at least one adequate trial of SRI medications or clomipramine and a course of CBT unless the participant is unable to access or tolerate CBT treatment.

   * In order to meet criteria for having had at least one adequate trial of SRI medication, participants must have been on a stable and minimal adequate dose of at least one SRI medication or clomipramine as defined by the literature for at least 12 weeks, and have a documented history of intolerable adverse effects at a higher dose as evaluated by the study psychiatrist and are therefore unable to increase the dose or complete the full 12 weeks, or have refused further SRI trials.

   Congruent with the literature, the range of minimally adequate doses to treat OCD are as follows: Clomipramine (Anafranil) 75-100 mg/day; Fluoxetine (Prozac) 20-60 mg/day; Paroxetine or Paroxetine CR (Paxil) 20-40 mg/day; Sertraline (Zoloft) 50-100 mg/day; Fluvoxamine (Luvox) 100-200 mg/day; Citalopram (Celexa) 20-40 mg; Escitalopram (Lexapro) 10-20 mg/day for a minimum of 12 weeks.
   * In order to meet criteria for having had an adequate course of CBT for OCD, patients should have received at least 8 sessions of Exposure and Response Prevention Therapy (EX/RP) by a licensed clinician trained in doing CBT for OCD. A CBT expert on our team will ensure that the clinician administering these exposures has had adequate training and experience in providing this treatment.
7. Participant is off all psychotropic and other types of drugs likely to interact with glutamate for at least 14 days before starting the study. The exceptions are SRI medications and short acting benzodiazepines for distressing anxiety or insomnia (which can be taken up to 24 hours prior to ketamine infusion). Participants will be off neuroleptics for 1 month and off fluoxetine for 6 weeks prior to the study.
8. For participants younger than 18, written informed assent by the participant and consent by the parent. For participants 19 and older, written consent by the participant and permission for legal guardian/parent to provide information.

Exclusion Criteria:

1. Family history of psychosis or substance abuse/dependence.
2. History of violence
3. Presence of psychotic symptoms or lifetime diagnosis of schizophrenia including any auditory or visual hallucinations or presence of delusional thinking, bipolar disorder, substance-induced psychotic disorder, psychosis due to general medical condition.
4. Severely depressed patients with the Children's Depression Rating Scale (CDRS) ≥ 60 or judged clinically to be at risk of suicide.
5. Current diagnosis of an eating disorder.
6. Current or past history of PTSD or significant trauma.
7. Current or past diagnosis of substance abuse/dependence.
8. Current or past diagnosis of pediatric autoimmune neuropsychiatric disorders associated with streptococcus (PANDAS). This will be defined by the following criteria: abrupt onset of OCD symptoms (often with comorbid tics) with a relapsing-remitting symptom course, a temporal association between symptom exacerbations and a Group-A beta-hemolytic streptococcal (GAS) infection, association with neurological abnormalities during exacerbations (adventitious movements, motoric hyperactivity, urinary hesitancy), and prepubertal age of onset.
9. Participants planning to commence cognitive-behavioral therapy during the period of the study or those who have begun CBT within 8 weeks prior to enrollment.
10. Documented history of hypersensitivity or intolerance to ketamine.
11. Female participants who are either pregnant or nursing or female participants of child bearing age who are sexually active and not taking hormonal birth control.
12. History of significant medical condition that might increase the risk of participation. This would include hypertension (BP > 140/90), chronic congestive heart failure, tachyarrhythmias, myocardial ischemia, intracranial mass lesions, head injury, globe injuries, or hydrocephalus.
13. Concurrent use of any medications that might increase the risk of participation. This would include: St. John's Wort, Tramadol or atracurium, due to potential adverse drug-drug interactions.
14. Positive urine screen for illicit drugs
15. Inability of participant or parent/guardian to read or understand English.
16. Documented history of adverse reaction to anesthesia.

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Goldberg, M.D., Principal Investigator — Columbia University/NYSPI
Locations (1):
- New York State Psychiatric Institute/Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rauch SL, Wedig MM, Wright CI, Martis B, McMullin KG, Shin LM, Cannistraro PA, Wilhelm S. Functional magnetic resonance imaging study of regional brain activation during implicit sequence learning in obsessive-compulsive disorder. Biol Psychiatry. 2007 Feb 1;61(3):330-6. doi: 10.1016/j.biopsych.2005.12.012. Epub 2006 Feb 21. PMID 16497278
- [Background] Atmaca M, Yildirim H, Ozdemir H, Tezcan E, Poyraz AK. Volumetric MRI study of key brain regions implicated in obsessive-compulsive disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jan 30;31(1):46-52. doi: 10.1016/j.pnpbp.2006.06.008. Epub 2006 Jul 20. PMID 16859819
- [Background] Graybiel AM, Rauch SL. Toward a neurobiology of obsessive-compulsive disorder. Neuron. 2000 Nov;28(2):343-7. doi: 10.1016/s0896-6273(00)00113-6. No abstract available. PMID 11144344
- [Background] Chakrabarty K, Bhattacharyya S, Christopher R, Khanna S. Glutamatergic dysfunction in OCD. Neuropsychopharmacology. 2005 Sep;30(9):1735-40. doi: 10.1038/sj.npp.1300733. PMID 15841109
- [Background] Rosenberg DR, MacMaster FP, Keshavan MS, Fitzgerald KD, Stewart CM, Moore GJ. Decrease in caudate glutamatergic concentrations in pediatric obsessive-compulsive disorder patients taking paroxetine. J Am Acad Child Adolesc Psychiatry. 2000 Sep;39(9):1096-103. doi: 10.1097/00004583-200009000-00008. PMID 10986805
- [Background] Rodriguez CI, Bender J Jr, Marcus SM, Snape M, Rynn M, Simpson HB. Minocycline augmentation of pharmacotherapy in obsessive-compulsive disorder: an open-label trial. J Clin Psychiatry. 2010 Sep;71(9):1247-9. doi: 10.4088/JCP.09l05805blu. PMID 20923629
- [Background] Coric V, Milanovic S, Wasylink S, Patel P, Malison R, Krystal JH. Beneficial effects of the antiglutamatergic agent riluzole in a patient diagnosed with obsessive-compulsive disorder and major depressive disorder. Psychopharmacology (Berl). 2003 May;167(2):219-20. doi: 10.1007/s00213-003-1396-z. Epub 2003 Mar 26. No abstract available. PMID 12658528
- [Background] Stewart SE, Jenike EA, Hezel DM, Stack DE, Dodman NH, Shuster L, Jenike MA. A single-blinded case-control study of memantine in severe obsessive-compulsive disorder. J Clin Psychopharmacol. 2010 Feb;30(1):34-9. doi: 10.1097/JCP.0b013e3181c856de. PMID 20075645
- [Background] Hezel DM, Beattie K, Stewart SE. Memantine as an augmenting agent for severe pediatric OCD. Am J Psychiatry. 2009 Feb;166(2):237. doi: 10.1176/appi.ajp.2008.08091427. No abstract available. PMID 19188297
- [Background] Rynn M, Puliafico A, Heleniak C, Rikhi P, Ghalib K, Vidair H. Advances in pharmacotherapy for pediatric anxiety disorders. Depress Anxiety. 2011 Jan;28(1):76-87. doi: 10.1002/da.20769. PMID 21225851
- [Background] Kararmaz A, Kaya S, Turhanoglu S, Ozyilmaz MA. Oral ketamine premedication can prevent emergence agitation in children after desflurane anaesthesia. Paediatr Anaesth. 2004 Jun;14(6):477-82. doi: 10.1111/j.1460-9592.2004.01224.x. PMID 15153210
- [Background] Dahmani S, Michelet D, Abback PS, Wood C, Brasher C, Nivoche Y, Mantz J. Ketamine for perioperative pain management in children: a meta-analysis of published studies. Paediatr Anaesth. 2011 Jun;21(6):636-52. doi: 10.1111/j.1460-9592.2011.03566.x. Epub 2011 Mar 29. PMID 21447047
- [Background] Finkel JC, Pestieau SR, Quezado ZM. Ketamine as an adjuvant for treatment of cancer pain in children and adolescents. J Pain. 2007 Jun;8(6):515-21. doi: 10.1016/j.jpain.2007.02.429. Epub 2007 Apr 16. PMID 17434801
- [Background] Rodriguez CI, Kegeles LS, Levinson A, Feng T, Marcus SM, Vermes D, Flood P, Simpson HB. Randomized controlled crossover trial of ketamine in obsessive-compulsive disorder: proof-of-concept. Neuropsychopharmacology. 2013 Nov;38(12):2475-83. doi: 10.1038/npp.2013.150. Epub 2013 Jun 19. PMID 23783065
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Marcus RJ, Victoria BA, Rushman SC, Thompson JP. Comparison of ketamine and morphine for analgesia after tonsillectomy in children. Br J Anaesth. 2000 Jun;84(6):739-42. doi: 10.1093/oxfordjournals.bja.a013585. PMID 10895748
- [Background] Aspinall RL, Mayor A. A prospective randomized controlled study of the efficacy of ketamine for postoperative pain relief in children after adenotonsillectomy. Paediatr Anaesth. 2001 May;11(3):333-6. doi: 10.1046/j.1460-9592.2001.00676.x. PMID 11359593
- [Background] Pediatric OCD Treatment Study (POTS) Team. Cognitive-behavior therapy, sertraline, and their combination for children and adolescents with obsessive-compulsive disorder: the Pediatric OCD Treatment Study (POTS) randomized controlled trial. JAMA. 2004 Oct 27;292(16):1969-76. doi: 10.1001/jama.292.16.1969. PMID 15507582
- [Background] Bloch MH, Landeros-Weisenberger A, Kelmendi B, Coric V, Bracken MB, Leckman JF. A systematic review: antipsychotic augmentation with treatment refractory obsessive-compulsive disorder. Mol Psychiatry. 2006 Jul;11(7):622-32. doi: 10.1038/sj.mp.4001823. Epub 2006 Apr 4. PMID 16585942
- [Background] Correll CU. Assessing and maximizing the safety and tolerability of antipsychotics used in the treatment of children and adolescents. J Clin Psychiatry. 2008;69 Suppl 4:26-36. PMID 18533766
- [Background] Papolos DF, Teicher MH, Faedda GL, Murphy P, Mattis S. Clinical experience using intranasal ketamine in the treatment of pediatric bipolar disorder/fear of harm phenotype. J Affect Disord. 2013 May;147(1-3):431-6. doi: 10.1016/j.jad.2012.08.040. Epub 2012 Nov 30. PMID 23200737
- [Derived] Ishimuro HS, Yanes-Lukin PK, Goldberg PH, Simpson HB, Rynn MA. Ketamine Treatment for Pediatric Refractory Obsessive: Five Open Label Cases. J Child Adolesc Psychopharmacol. 2025 Apr;35(3):167-170. doi: 10.1089/cap.2024.0127. Epub 2025 Feb 3. PMID 39899368

RESULTS

PARTICIPANT FLOW:
Groups:
- Adolescent OCD Ketamine Group: Open trial of ketamine IV for adolescents with treatment refractory OCD
Period: Overall Study
Arm/Group | Adolescent OCD Ketamine Group
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Demographics: Demographics of participants
Arm/Group | Demographics
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (1.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Description: The CY-BOCS is a semi-structured measure of OCD severity with excellent inter-rater reliability, internal consistency, and test-retest reliability. It is validated in those starting at age 7 and used in studies up to age 20. The CYBOCS differs from the adult YBOCS only in its use of simpler language. The CY-BOCS consists of 10 items which are summed up to derive the total CY-BOCS score. The total score ranges from 0-40 with higher scores indicating greater severity of OCD symptoms.
Time Frame: Screening, Baseline, Day 7, Day 17, 3-Month; Baseline and Day 14 pre-specified to be reported
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ketamine Treatment Group: Adolescents and young adults with OCD who received an intravenous ketamine infusion.
Arm/Group | Ketamine Treatment Group
Number analyzed (Participants) | 5
score on a scale
  CY-BOCS Baseline | 29.00 (5.52)
  CY-BOCS Day 14 | 26.20 (5.59)
Statistical Analysis 1: Comparison: Ketamine Treatment Group; Paired sample t-test was calculated to test mean difference between CY-BOCS scores at the time points Baseline and Day 14; Test type: Superiority; p = .20, t-test, 2 sided; Mean Difference (Final Values) = 1.53, 95% CI 2-sided [-2.27 to 7.87], Standard Error of Mean 1.83

2. Primary Outcome: Clinical Global Impressions - Severity Scale (CGI-S)
Description: The CGI-S is a clinician rated 7-point rating scale for the severity of a participant's illness relative to the clinician's experience of working with this particular population. The score ranges from 1-7 with higher scores indicating greater illness severity.
Time Frame: Screening, Baseline, Day 7, Day 17, 3-Month; Baseline and Day 14 pre-specified to be reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Treatment Group
Number analyzed (Participants) | 5
score on a scale
  CGI-S Baseline | 5.80 (0.45)
  CGI-S Day 14 | 5.00 (1.00)
Statistical Analysis 1: Comparison: Ketamine Treatment Group; Paired sample t-test was calculated to test mean difference between CGI-S scores at the time points Baseline and Day 14; Test type: Superiority; p = .18, t-test, 2 sided; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [-.56 to 2.16], Standard Error of Mean .49

3. Secondary Outcome: OCD Visual Analogue Scale (OCD-VAS)
Description: The OCD-VAS is a one-item unipolar scale to assess OCD symptoms over a rapid time frame ("No obsessions" to "Constant obsessions"). The scale ranges from 0-10 with higher scores indicating higher presence of obsessions.
Time Frame: Screening, Baseline, Day 1-14, 3-Month; Baseline and Day 14 pre-specified to be reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Treatment Group
Number analyzed (Participants) | 5
score on a scale
  OCD-VAS Baseline | 5.00 (1.00)
  OCD-VAS Day 14 | 5.00 (2.12)
Statistical Analysis 1: Comparison: Ketamine Treatment Group; Paired sample t-test was calculated to test mean difference between OCD-VAS scores at the time points Baseline and Day 14; Test type: Superiority; p = 1.00, t-test, 2 sided; Mean Difference (Final Values) = .00, 95% CI 2-sided [-2.78 to 2.78], Standard Error of Mean 1.00

4. Secondary Outcome: Yale-Brown Obsessive Compulsive Challenge Scale (Y-BOCCS)
Description: The Y-BOCCS is self-report scale which assesses OCD symptoms on a 5-point likert scale ("None" to "Extreme"). It consists of 10 items which are summed up to derive the total Y-BOCCS score. The total score ranges from 0-40 with higher scores indicating higher prevalence of OCD symptoms.
Time Frame: Screening, Baseline, Day 1-14, 3-Month; Baseline and Day 14 pre-specified to be reported
Population: One participant was missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Treatment Group
Number analyzed (Participants) | 4
score on a scale
  Y-BOCCS Baseline | 18.25 (7.27)
  Y-BOCCS Day 14 | 16.50 (5.32)
Statistical Analysis 1: Comparison: Ketamine Treatment Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .77, t-test, 2 sided; Mean Difference (Final Values) = .32, 95% CI 2-sided [-15.46 to 18.96], Standard Error of Mean 5.41

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the ketamine infusion and for two hours post-infusion. Following the infusion, adverse events were assessed daily for a period of 14 days and at a 3-month follow-up visit.
Arm/Group | Ketamine Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Treatment Group (N=5)
Psychiatric Hospitalization (Psychiatric disorders) | 1 (1) — Hospitalization for 5 days due to worsening depression and passive suicidal ideation two months after the ketamine infusion. This was not thought to be related directly to the ketamine infusion. IRB was informed.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Treatment Group (N=5)
Dissociation (Psychiatric disorders) | 4 (4) — Mild dissociation during the ketamine infusion.
Dizziness (Nervous system disorders) | 2 (2) — Dizziness during ketamine infusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT02422290/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT02422290/SAP_001.pdf